CLINICAL TRIAL: NCT01143753
Title: An Open-Label, Multiple Ascending Dose (MAD) Study of the Selective BRAF Inhibitor RO5212054 (PLX3603) to Evaluate Safety, Tolerability and Pharmacokinetics in Patients With BRAF V600-Mutated Advanced Solid Tumours
Brief Title: A Study of RO5212054 (PLX3603) in Participants With BRAF V600-Mutated Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP25247; 2010-018330-42 (EudraCT Number)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- RO5212054: Continuous Dosing Cohort (Experimental): Participants will receive RO5212054 in escalating dose levels.
  Interventions: Drug: RO5212054
- RO5212054: New Formulation (F05) Bridging Cohort (Experimental): Participants will receive RO5212054 as a single dose of new formulation (F05-150 mg film-coated tablet with different ratios of ingredients than F03 to increase bioavailability) and a single dose of current clinical Formulation (F03-150 mg film-coated tablet) in a cross-over manner. Participants will be alternately assigned to receive either F05 or F03 as their first dose, followed by the opposite Formulation as their second dose. Dose of RO5212054 will be decided based on the results of continuous dosing cohort.
  Interventions: Drug: RO5212054

INTERVENTIONS:
Drug: RO5212054 — Participants will receive RO5212054 at a starting dose of 200 milligrams (mg) orally once daily in each 21 day cycle. Dose levels for escalation will be decided based on the safety assessment of previous cohort. Dose escalations in increments of 50-100 percent are planned.
  Other Names: PLX3603

SUMMARY:
This open-label, multi-center study will evaluate the safety, tolerability, and pharmacokinetics of RO5212054 [PLX3603] in participants with BRAF V600-mutated advanced solid tumors. Cohorts of participants will receive escalating oral doses of RO5212054. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Dose-escalation phase: Histologically confirmed, newly diagnosed or relapsed/ refractory unresectable American Joint Committee on Cancer (AJCC) Stage IIIC or IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate liver, renal and bone marrow function

Exclusion Criteria:

* Participants for whom standard therapy exists and is considered appropriate by the investigator
* Prior treatment with an inhibitor of BRAF (sorafenib allowed)
* Active Central nervous system (CNS) lesions, or history of or known carcinomatous meningitis
* Treatment with any chemotherapy, radiotherapy, immunotherapy or investigational agent within 28 days prior to first dose of study drug
* Anticipated or ongoing anti-cancer therapies other than those administered in this study
* Serious cardiovascular illness within the 6 months prior to study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-07-27 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicity | Baseline up to 21 days
Maximal Tolerated Dose of RO5212054 | Baseline up to 21 days
Maximum Plasma Concentration of RO5212054 | Baseline up to cycle 10 (cycle length: 21 days) (detailed timeframe is given in description)
  Detailed timeframe:
  Pre-dose (0 hour [hr]): Day 1 of Cycles 1-10; Days 4, 8, 15 of Cycle 1. Post-dose: 1, 2, 4, 8, 12, 24 hr on Day 1 Cycle 1; Between 2-4 hr (1 sample) on Day 8 Cycle 1 and Day 1 Cycles 2-9; 1, 2, 4, 8, Between 10-12 hr (1 sample), 24 hr on Day 15 Cycle 1 (cycle length: 21 days)
Time to Reach Maximum Plasma Concentration of RO5212054 | Baseline up to cycle 10 (cycle length: 21 days) (detailed timeframe is given in description)
  Detailed timeframe:
  Pre-dose (0 hr): Day 1 of Cycles 1-10; Days 4, 8, 15 of Cycle 1. Post-dose: 1, 2, 4, 8, 12, 24 hr on Day 1 Cycle 1; Between 2-4 hr (1 sample) on Day 8 Cycle 1 and Day 1 Cycles 2-9; 1, 2, 4, 8, Between 10-12 hr (1 sample), 24 hr on Day 15 Cycle 1 (cycle length: 21 days)
Area Under The Plasma Concentration-Time Curve of RO5212054 | Baseline up to cycle 10 (cycle length: 21 days) (detailed timeframe is given in description)
  Detailed timeframe:
  Pre-dose (0 hr): Day 1 of Cycles 1-10; Days 4, 8, 15 of Cycle 1. Post-dose: 1, 2, 4, 8, 12, 24 hr on Day 1 Cycle 1; Between 2-4 hr (1 sample) on Day 8 Cycle 1 and Day 1 Cycles 2-9; 1, 2, 4, 8, Between 10-12 hr (1 sample), 24 hr on Day 15 Cycle 1 (cycle length: 21 days)

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to approximately 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Australia (3):
  - Royal Adelaide Hospital; Oncology, Adelaide, South Australia
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
  - Royal Melbourne Hospital; Hematology and Medical Oncology, Parkville, Victoria
- Rigshospitalet, Onkologisk Klinik, København Ø, Denmark
- Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona, Spain

REFERENCES:
- [Derived] Dienstmann R, Lassen U, Cebon J, Desai J, Brown MP, Evers S, Su F, Zhang W, Boisserie F, Lestini B, Schostack K, Meresse V, Tabernero J. First-in-Man Dose-Escalation Study of the Selective BRAF Inhibitor RG7256 in Patients with BRAF V600-Mutated Advanced Solid Tumors. Target Oncol. 2016 Apr;11(2):149-56. doi: 10.1007/s11523-015-0381-x. PMID 26310975